CLINICAL TRIAL: NCT00014950
Title: Pulmonary Benefits of Cystic Fibrosis Neonatal Screening
Brief Title: Benefits and Risks of Newborn Screening for Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Single Group | Purpose: Diagnostic
Other Study IDs: Farrell (completed); R01DK034108 (NIH); GCRC
Record Dates: First submitted 2001-04-14; First posted 2001-04-16 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Cystic Fibrosis; Lung Disease; Pseudomonas Infections
Keywords: Cystic Fibrosis; Immunoreactive trypsinogen; deltaF508- CFTR gene; newborn screening; Pseudomonas aeruginosa infection; nutrition; pulmonary status; meconium ileus; growth; Genetic counseling; risk communication
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases; Pseudomonas Infections; Meconium Ileus

INTERVENTIONS:
Procedure: CF newborn screening

SUMMARY:
Although cystic fibrosis (CF) is the most common, life-threatening autosomal recessive genetic disorder of the white population, there are often delays in diagnosis and hence start of treatment. Advances of the past two decades have made CF screening feasible using routinely collected neonatal blood specimens and measuring an enzyme level followed by CF mutation DNA analysis. Our overall goal of the study is to see if early diagnosis of CF through neonatal screening will be medically beneficial without major risks. ''Medically beneficial'' refers to better nutrition and/or pulmonary status, whereas '' risks'' include laboratory errors, miscommunication or misunderstanding, and adverse psychosocial consequences. Specific aims include assessment of the benefits, risks, costs, quality of life, and cognitive function associated with CF neonatal screening and a better understanding of the epidemiology of CF.

A comprehensive, randomized clinical trial emphasizing early diagnosis as the key variable has been underway since 1985. Nutritional status has been assessed using height and weight measurements and biochemical methods. The results have demonstrated significant benefits in the screened (early diagnosis) group. We are now focusing on the effect of early diagnosis of CF on pulmonary outcome. Pulmonary status is measured using chest radiographs, chest scans using high resolution computerized tomography, and pulmonary function tests. Other factors that we are looking at include risk factors for the acquisition of respiratory pathogens such as Pseudomonas aeruginosa, quality of life and cognitive function of children with CF who underwent early versus delayed diagnosis, as well as the cost effectiveness of screening and the costs of diagnosis and treatment of CF throughout childhood.

If the questions underlying this study are answered favorably, it is likely that neonatal screening using a combination of enzyme level (immunoreactive trypsinogen) and DNA test will become the routine method for identifying new cases of CF not only in the State of Wisconsin, but throughout the country.

ELIGIBILITY:
Inclusion Criteria:

* Must have been born in the State of Wisconsin
* Must have been born between April 15, 1985 and June 30, 1994
* Must have had a valid newborn screening test for cystic fibrosis in the first 28 days of life.
* Must have a sweat chloride test greater or equal to 60 mmol/Liter
* Parental consent

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Philip M. Farrell, MD, PhD, Principal Investigator — Dean University of Wisconsin Medical School; Michael J. Rock, M.D. — Dept. Pediatrics, UW Hospital; Mark Splaingard — Children's Hospital and Health System Foundation, Wisconsin; Anita Laxova — Dept. Pediatrics, UW Madison
Locations (2):
- United States (2):
  - University of Wisconsin, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Crossley JR, Elliott RB, Smith PA. Dried-blood spot screening for cystic fibrosis in the newborn. Lancet. 1979 Mar 3;1(8114):472-4. doi: 10.1016/s0140-6736(79)90825-0. PMID 85057
- [Background] Neonatal screening for cystic fibrosis: position paper. Pediatrics. 1983 Nov;72(5):741-5. No abstract available. PMID 6634283
- [Background] Fost N, Farrell PM. A prospective randomized trial of early diagnosis and treatment of cystic fibrosis: a unique ethical dilemma. Clin Res. 1989 Sep;37(3):495-500. No abstract available. PMID 2673641
- [Background] Farrell PM, Kosorok MR, Laxova A, Shen G, Koscik RE, Bruns WT, Splaingard M, Mischler EH. Nutritional benefits of neonatal screening for cystic fibrosis. Wisconsin Cystic Fibrosis Neonatal Screening Study Group. N Engl J Med. 1997 Oct 2;337(14):963-9. doi: 10.1056/NEJM199710023371403. PMID 9395429
- [Background] Farrell PM. Improving the health of patients with cystic fibrosis through newborn screening. Wisconsin Cystic Fibrosis Neonatal Screening Study Group. Adv Pediatr. 2000;47:79-115. No abstract available. PMID 10959441
- [Background] Farrell PM, Kosorok MR, Rock MJ, Laxova A, Zeng L, Lai HC, Hoffman G, Laessig RH, Splaingard ML. Early diagnosis of cystic fibrosis through neonatal screening prevents severe malnutrition and improves long-term growth. Wisconsin Cystic Fibrosis Neonatal Screening Study Group. Pediatrics. 2001 Jan;107(1):1-13. doi: 10.1542/peds.107.1.1. PMID 11134427